CLINICAL TRIAL: NCT05546697
Title: COMPARE: Comparing Behavior Therapy and Yoga for Treating Depression Among Adults
Brief Title: Comparing Behavior Therapy and Yoga for Treating Depression Among Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Butler Hospital (Other); Hennepin Healthcare Research Institute (Other); Medical University of South Carolina (Other); Brown University (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Louisa Grandin Sylvia, Associate Director, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022P001701
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Depression
Keywords: Yoga-based Intervention; Behavioral Activation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga-based Intervention (Active Comparator): Yoga classes will be gentle and physically accessible for people who are naïve to yoga. Teachers will frequently guide participants to focus on their breathing and coordinate movements with breath. Teachers will offer variations on the postures and encourage participants to choose variations that provide some challenge but do not cause strain or pain. Classes will be 1 hour long and include a brief sitting meditation, warm-ups, standing postures, and a final resting meditation. All participants will be invited to attend a synchronous yoga class via a HIPAA-compliant videoconference option once per week during the first 3 months of the study. Classes will be offered at multiple times throughout the week.
  Interventions: Other: Online- Yoga-based Intervetion
- Behavioral Activation (Active Comparator): The goal of Behavioral Activation Psychotherapy is to help people identify and (re)engage in meaningful and positive activities through psychoeducation, identification of values and associated activities, goal setting, problem-solving, and monitoring of goal completion. There will be a BA manual for therapists and training provided by study staff on the manual (e.g., asynchronous and synchronous training sessions). BA therapists will be community clinicians. BA will be provided individually via telehealth and will be billed to participant insurance. At the start of BA treatment, participants will be oriented to the time-limited nature of BA, with the expectation that they will attend 8 sessions over the course of 3 months.
  Interventions: Behavioral: Online- BA

INTERVENTIONS:
Other: Online- Yoga-based Intervetion — See arms description
  Arms: Yoga-based Intervention
Behavioral: Online- BA — See arms description
  Arms: Behavioral Activation

SUMMARY:
This is a parallel group study design. The investigators propose to compare an online, synchronous group-based yoga intervention developed for individuals with depression to an online, synchronous individualized, evidence-based behavioral therapy for depression, or Brief Behavioral Activation Treatment for Depression (BA). This study is a multi-site randomized trial of adults with clinically significant depressive symptoms. Participants (N=518) will be randomized in an equal allocation ratio (i.e., 1:1) across two intervention groups: yoga and BA. Interventions will be provided over a 12-week period and assessments will occur at baseline (week 0), week 6, week 12, week 18, and week 24.

DETAILED DESCRIPTION:
The first goal of the proposed research is to determine whether a hatha yoga program for depression is non-inferior to BA in reducing depressive symptoms over a 6-month period.

Our second goal is to identify individual-level characteristics that predict heterogeneity of treatment effect (HTE) to develop guidance for matching patients to the optimal depression treatment.

Sample- Our sample will be representative of the target population: individuals with depression. There are several aspects of the current study design that the investigators believe will enhance recruitment in diverse patient populations.

* Both study interventions will be offered via telehealth to reduce barriers to access (e.g., childcare, time, parking/transportation costs, less time out of work).
* The investigators have study funds to cover the costs of the technology for people who do not have a device or home-based internet access. Further, to decrease barriers related to digital literacy, study staff will be proactive about assisting participants with setting up technology, using technology and troubleshooting if needed.
* The investigators have study funds to pay for the BA therapists for participants who are uninsured.
* The investigators have study funds to offer the yoga intervention free of charge to participants.
* The investigators will offer study participation to Spanish-speakers.
* The investigators have an Advisory Board of stakeholders with diverse backgrounds (i.e., racially and ethnically diverse as well as diversity in socioeconomic status, educational background, and clinical features) to assist with the implementation and oversight of this study.

Participants will be paid for completing study assessments, they will not be compensated for attending study intervention sessions.

Assessments occur at Baseline (week 0, prior to randomization), and weeks 6, 12, 18, and 24. All self-report assessments will be available in English or Spanish. When an assessment is due, participants will be sent an automated link to complete the assessments via REDCap. In addition, they will receive reminders if they do not complete the assessment, and, if needed, follow-up phone calls from study staff. It is expected that the assessments at Weeks 0 (baseline) and 24 (end of treatment) will take approximately 45 min to complete, at Week 12 will take approximately 30 min to complete and at Weeks 6 and 18 will take approximately 20 min to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years old or older
2. Depressive symptoms at study entry (PHQ-9≥10)
3. Provides informed consent
4. Able to read and understand English or Spanish.
5. Live in NC, MA, MN, or RI
6. Has a healthcare provider (a primary care provider, clinic, or mental health care provider) whom the participant could contact if medical care were needed

Exclusion Criteria:

1. PHQ-9 > 20
2. A bone fracture or joint surgery in the past 6 months
3. Unable to walk
4. Severe heart failure or lung disease
5. Had a healthcare provider tell them it is unsafe to exercise
6. Currently pregnant
7. Are already engaged in study interventions (i.e., engaged in yoga practice or psychotherapy more than once in the past 4 weeks or has an intake scheduled for psychotherapy in the next 4 weeks).
8. Have active suicidal thinking (i.e., PHQ-9 item 9 ≥1 and a positive response to CSSR-S screener items 3, 4, 5, or 6 [Past 3 months])
9. Are currently experiencing manic symptoms (Altman Self-Rating Mania Scale score ≥ 6)
10. Unable to complete study procedures (i.e., attend yoga classes, BA sessions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Week: 0
  It is a 9-item self-report questionnaire that is widely used to assess depression symptom severity. A PHQ-9 score ≥10 has a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.
Patient Health Questionnaire-9 (PHQ-9) | Week: 6
  It is a 9-item self-report questionnaire that is widely used to assess depression symptom severity. A PHQ-9 score ≥10 has a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.
Patient Health Questionnaire-9 (PHQ-9) | Week:12
  It is a 9-item self-report questionnaire that is widely used to assess depression symptom severity. A PHQ-9 score ≥10 has a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.
Patient Health Questionnaire-9 (PHQ-9) | Week:18
  It is a 9-item self-report questionnaire that is widely used to assess depression symptom severity. A PHQ-9 score ≥10 has a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.
Patient Health Questionnaire-9 (PHQ-9) | Week: 24
  It is a 9-item self-report questionnaire that is widely used to assess depression symptom severity. A PHQ-9 score ≥10 has a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.

SECONDARY OUTCOMES:
World Health Organization-5 Well-Being Index (WHO-5) | Week: 0, 6, 12, 18, 24
  It is a 5-item self-report questionnaire with positively-worded statements related to positive mood, vitality, and general interest over the prior two weeks. The WHO-5 is reliable, has shown strong construct validity as a measure of general quality of life, and is sensitive to change.
PROMIS-29 Anxiety Subscale | Week: 0, 6, 12, 18, 24
  Part of the PROMIS-29 scale which has seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, social functioning, sleep disturbance) with four items in this domain. PROMIS scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe anxiety, respectively. It has demonstrated good psychometric properties.
PROMIS-29 Sleep Subscale | Week: 0, 6, 12, 18, 24
  Part of the PROMIS-29 scale which has seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, social functioning, sleep disturbance) with four items in this domain. PROMIS scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe sleep disturbance respectively. It has demonstrated good psychometric properties.

OTHER OUTCOMES:
PROMIS Anger | Week: 0, 6, 12, 18, 24
  It is a 5-item self-report scale used to assess the exploratory outcome of irritability. PROMIS scores of 5, 10, 15, 20, and 25 represented minimal, mild, moderate, moderately severe, and severe anger, respectively.
PROMIS-29 Physical Functioning Subscale | Week: 0, 6, 12, 18, 24
  Part of the PROMIS-29 scale which has seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, social functioning, sleep disturbance) with four items in this domain. PROMIS scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe physical function, respectively. It has demonstrated good psychometric properties.
PROMIS-29 Social Functioning Subscale | Week: 0, 6, 12, 18, 24
  Part of the PROMIS-29 scale which has seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, social functioning, sleep disturbance) with four items in this domain. PHQ-9 scores of 5, 10, 15, and 20 represented severe, moderately severe, moderate, and mild physical functioning, respectively. It has demonstrated good psychometric properties.
PROMIS-29 Pain Interference | Week: 0, 6, 12, 18, 24
  Part of the PROMIS-29 scale which has seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, social functioning, sleep disturbance) with four items in this domain. PROMIS scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe pain interference, respectively. It has demonstrated good psychometric properties.

CONTACTS AND LOCATIONS:
Overall Officials: Louisa Sylvia, PhD, Principal Investigator — Massachusetts General Hospital; Lisa Uebelacker, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Giuliana Chau, Boston, Massachusetts, United States